CLINICAL TRIAL: NCT05833334
Title: Co-developing and Pilot Testing a Risk-tailored, Technology-supported Intervention to Increase Home Radon Testing in New Hampshire and Vermont
Brief Title: Healthy Homes Study
Acronym: HHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Judith R. Rees, Associate Professor, Epidemiology; Associate Professor, Community & Family Medicine; Associate Director, Community Outreach and Engagement, Dartmouth Cancer Center, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02001931; NCI-2024-01233 (Other: NCI)
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Home Air Radon Testing; Lung Cancer
Keywords: Radon testing; Behavior change; Smoking; Air quality
MeSH Terms: conditions — Lung Neoplasms; Smoking | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Public health infographic (AIM 3) (Active Comparator): Participants will view a standard public health infographic about home air radon testing and will receive information about requesting a free home air radon test kit from their state radon program.
  Interventions: Behavioral: Public health infographic (AIM 3)
- Online health promotion intervention tailored by smoking status (AIM 3) (Experimental): Participants will view an online health promotion intervention about home air radon testing, with messaging tailored based on whether the participant smokes or does not smoke. Participants will also receive information about requesting a free home air radon test kit from their state radon program.
  Interventions: Behavioral: Online health promotion intervention tailored by smoking status (AIM 3)
- Online health promotion intervention tailored by smoking status, plus reminder messages (AIM 3) (Experimental): Participants will view an online health promotion intervention about home air radon testing, with messaging tailored based on whether the participant smokes or does not smoke. Participants will also receive information about requesting a free home air radon test kit from their state radon program, as well as reminder messages about radon testing for about two months after initially viewing the online intervention component.
  Interventions: Behavioral: Online health promotion intervention tailored by smoking status, plus reminder messages (AIM 3)
- Focus group with educational overview (AIM 1) (Experimental): Participants will participate in a focus group discussion about radon testing and will receive a brief educational overview about radon testing.
  Interventions: Behavioral: Focus group with educational overview (AIM 1)

INTERVENTIONS:
Behavioral: Public health infographic (AIM 3) — Standard public health infographic about home air radon testing, plus information about requesting a free home air radon test kit
  Arms: Public health infographic (AIM 3)
Behavioral: Online health promotion intervention tailored by smoking status (AIM 3) — Online health promotion intervention with messaging about home air radon testing tailored by the participant's stated smoking status, plus information about requesting a free home air radon test kit
  Arms: Online health promotion intervention tailored by smoking status (AIM 3)
Behavioral: Online health promotion intervention tailored by smoking status, plus reminder messages (AIM 3) — Online health promotion intervention with messaging about home air radon testing tailored by the participant's stated smoking status, plus information about requesting a free home air radon test kit, plus reminder messages about home air radon testing sent over two months
  Arms: Online health promotion intervention tailored by smoking status, plus reminder messages (AIM 3)
Behavioral: Focus group with educational overview (AIM 1) — 90-minute online focus group discussion about home air radon testing, plus an educational overview about home air radon testing using a standard public health infographic
  Arms: Focus group with educational overview (AIM 1)

SUMMARY:
This study is about home air radon testing and has two phases.

The goal of the first phase is to learn about renters' and homeowners' views and plans related to radon testing. The main question this phase aims to answer is:

1. Does taking part in a focus group with information about radon testing change people's plans to test for radon?

Participants in the first study phase will:

* Take a survey about their views on and plans for radon testing.
* Take part in a focus group discussion about radon testing, during which they will receive information about radon testing.
* Right after the focus group, take a survey about their plans for radon testing.

The second phase is a pilot interventional study. The goal is to test interventions about radon testing with renters and homeowners who smoke and do not smoke. The main questions this phase aims to answer are:

1. Does the recruitment strategy result in enough participants enrolling within 3 months?
2. Will at least 80% of participants complete data collection activities?
3. Will more participants who view an online intervention developed by the researchers request free radon test kits, set them up in their homes, and complete radon testing, compared to participants who view a standard public health infographic? And will even more participants who receive reminder messages, in addition to the online intervention, request free radon test kits, set them up in their homes, and complete radon testing?

Participants in this second phase will:

* Take a survey about their views on and plans for radon testing.
* View an intervention about radon testing.
* Right after viewing the intervention, take a survey about their views on and plans for radon testing.
* 2 months later, take a survey about what, if any, steps they've taken to test their homes for radon.
* Provide the researchers permission to collect data from their State Radon Program on: a) whether they requested a free radon test kit and b) whether testing was completed.

Some participants will receive reminder messages for 2 months after viewing the intervention.

Researchers will compare an online intervention they developed about radon testing to: a) a standard public health infographic and b) their online intervention combined with reminder messages about radon testing. They will compare the interventions by proportion of participants who: a) request a free radon test kit from their State Radon Programs, b) set-up the radon test kit in their homes, and c) complete radon testing.

DETAILED DESCRIPTION:
This study is a pilot research study.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have a valid mailing address in New Hampshire or Vermont,
* Have not tested their current homes for radon,
* Rent or own their home, and
* Live at their home year-round

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-08-24 (Estimated); Study Completion 2027-08-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled in the study (AIM 3) | 3 months
  Number of participants who consent into the study and meet eligibility criteria within 3 months of study opening to enrollment.
Proportion of study participants who complete all study surveys (AIM 3) | 2 months
  Proportion of study participants who complete all study-related surveys, including the pre-intervention survey, post-intervention survey, and follow-up survey at 2 months post-intervention.
Proportion of participants who request a home radon test kit at 18 months (AIM 3) | 18 months
  Proportion of participants, by study arm, who request a free home radon test kit from the New Hampshire Radon Program or Vermont Radon Program in the 18 months following the intervention, the New Hampshire Radon Program or Vermont Radon Program, as reported by the state radon programs; radon test kits are attributed to participants if the state radon program records match the participant's name and/or address of home residence.
Proportion of participants who request a home radon test kit at 2 months (AIM 3) | 2 months
  Proportion of participants, by study arm, who request a free home radon test kit from the New Hampshire Radon Program or Vermont Radon Program in the 18 months following the intervention, the New Hampshire Radon Program or Vermont Radon Program, as reported by the state radon programs; radon test kits are attributed to participants if the state radon program records match the participant's name and/or address of home residence.
Proportion of participants who set-up a home radon test kit in their home (AIM 3) | 2 months
  Proportion of participants, by study arm, who report setting up the a home radon test kit in their home at two months post-intervention.
Proportion of participants who complete home radon testing at 18 months (AIM 3) | 18 months
  Proportion of participants, by study arm who either: a) report completing radon testing via the follow-up survey at two months post-intervention, or b) submit a home radon test kit for analysis through the New Hampshire Radon Program or Vermont Radon Program, as reported by the state radon programs; radon test kits are attributed to participants if the state radon program records match the participant's name and/or address of home residence.
Proportion of participants who complete home radon testing at 2 months (AIM 3) | 2 months
  Proportion of participants, by study arm who either: a) report completing radon testing via the follow-up survey at two months post-intervention, or b) submit a home radon test kit for analysis through the New Hampshire Radon Program or Vermont Radon Program, as reported by the state radon programs; radon test kits are attributed to participants if the state radon program records match the participant's name and/or address of home residence.

SECONDARY OUTCOMES:
Change in participants' intentions to test the air in their homes for radon in the next 12 months (AIM 1) | Baseline (pre-test, approximately 1-4 weeks before intervention), immediately after the intervention (post-test)
  Intention to test will be measured on a scale of 0 to 10, with 0 indicating they definitely will not test their home air for radon and 10 indicating they definitely will test their home air for radon in the next 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Rees, BM, BCh, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Rian M Hasson, MD, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No